CLINICAL TRIAL: NCT05665517
Title: User Evaluation of a Chat-based Instant Messaging Support Health Education Program for Chronic Kidney Disease: Effectiveness and Gender Differences
Brief Title: Chat-based Instant Messaging Support Health Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Jong-Long Guo, Distinguished Professor, National Taiwan Normal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 109-E-04
Record Dates: First submitted 2022-09-22; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Chatbot; Push notification; Users' evaluation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: At the first meeting, the participants completed the pre-test of the CKD patient's simple health literacy evaluation and were invited to use the "Chatbot Little K Nurse", which was an intervention of CKD chat-based instant messaging support health education system.
  After the first week, the first System Usability Scale (SUS) measurement was completed, whereas the second SUS measurement was completed in the fourth week. After completing the intervention in the 12th week, the participant's health literacy was reassessed through a post-test, and the third SUS assessment was performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chatbot Little K Nurse (Experimental): The CKD chat-based instant messaging support health education system in this study was named "Chatbot Little K Nurse" and connected to the Line platform to set up a one-to-one line. K stands for "kidney." Each group contained three parties: patients with CKD (participants ), Chatbot Little K Nurse (virtual), and an instructor (health teacher) for an enhanced intervention. According to the handbook of CKD health management by the Health Promotion Administration (2018b) and the CKD Clinical Diagnosis and Treatment Guidelines for literature investigation in Taiwan, 350 groups of question-and-answer (Q&A) corpora were formed.
  Interventions: Device: Chatbot Little K Nurse

INTERVENTIONS:
Device: Chatbot Little K Nurse — The CKD chat-based instant messaging support health education system in this study was named "Chatbot Little K Nurse" and connected to the Line platform to set up a one-to-one line. K stands for "kidney." Each group contained three parties: patients with CKD (participants ), Chatbot Little K Nurse (virtual), and an instructor (health teacher) for an enhanced intervention. According to the handbook of CKD health management by the Health Promotion Administration (2018b) and the CKD Clinical Diagnosis and Treatment Guidelines for literature investigation in Taiwan, 350 groups of question-and-answer (Q&A) corpora were formed.

SUMMARY:
The purpose of this study is to explore the effectiveness of a CKD-specific chatbot-based instant messaging support health education (CIM-SHE) program and determine its user evaluation by CKD patients.

A pre- and post-study design was employed and 60 patients were invited to join a three-month program for chronic kidney disease health education; 55 successfully completed the intervention. Data were collected from April to November, 2020, using a structured questionnaire. Paired t-tests and generalized equation estimation were used to examine the intervention effectiveness and users' evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. adults over 20 years old
2. diagnosed chronic kidney disease
3. the ability to operate technologies
4. intact cognition

Exclusion Criteria:

Who was undergoing kidney dialysis, unconsciousness, dementia, or any other mental illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Chronic kidney disease subjects' health literacy and disease knowledge | 12 weeks
  A chronic kidney disease specific health literacy and knowledge assessment tool consists of two parts: (1) chronic kidney disease specific health literacy (communicative literacy) and (2) disease knowledge. Participants scored one point for each correct answer and 0 points for wrong answers. A paired sample t-test was used to analyze chronic kidney disease subjects' health literacy (pre-test vs. post-test).
System usability scale was developed to subjectively evaluate the user's operating system to understand and ensure its usability and quality. | 12 weeks
  The System usability scale consisted of 10 items rated on a Likert-type scale ranging from one (strongly disagree) to five (strongly agree). In this study, items 1-5 and 6-10 were considered positive and negative, respectively. For positive items, we subtracted 1 point and for negative items, we subtracted 5 points from the score of the items. The generalized estimating equation was used to evaluate the change of System usability scale scores at three time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Long Guo, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University,, Taipei, Taiwan

REFERENCES:
- [Derived] Chen NJ, Huang CM, Fan CC, Lu LT, Lin FH, Liao JY, Guo JL. User Evaluation of a Chat-Based Instant Messaging Support Health Education Program for Patients With Chronic Kidney Disease: Preliminary Findings of a Formative Study. JMIR Form Res. 2023 Sep 19;7:e45484. doi: 10.2196/45484. PMID 37725429